CLINICAL TRIAL: NCT03978442
Title: CPT-SMART for Treatment of PTSD and Cigarette Smoking
Acronym: CPT-SMART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHBB-008-18F
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Smoking; Stress Disorders, Post-Traumatic
Keywords: Stress Disorders, Post-Traumatic; Smoking
MeSH Terms: conditions — Smoking; Stress Disorders, Post-Traumatic | interventions — Bupropion; 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Intervention Model Description: Randomized, two-arm clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CPT-SMART (Experimental): COGNITIVE PROCESSING THERAPY with SMOKING ABSTINENCE REINFORCEMENT THERAPY (CPT-SMART) - an intervention that combines evidence-based PTSD treatment with guideline-concordant cognitive-behavioral smoking cessation counseling, bupropion, and intensive behavioral therapy through CM.
  Interventions: Behavioral: Smoking Cessation Cognitive Behavioral Therapy (CBT); Drug: Bupropion; Behavioral: Cognitive Processing Therapy; Behavioral: Smoking Abstinence Reinforcement Therapy
- Combined Contact Yoked Control (Active Comparator): COMBINED CONTACT YOKED CONTROL (CCYC) - an intervention that is identical to CPT-SMART for PTSD and smoking treatment, except for using non-contingent payment (i.e., yoked CM) to control for compensation and monitoring.
  Interventions: Behavioral: Smoking Cessation Cognitive Behavioral Therapy (CBT); Drug: Bupropion; Behavioral: Cognitive Processing Therapy; Behavioral: Yoked Contingency Management

INTERVENTIONS:
Behavioral: Smoking Cessation Cognitive Behavioral Therapy (CBT) — 12 sessions of cognitive behavioral therapy for smoking cessation, designed to help participants prepare for quitting smoking, make a quit attempt, and stay quit from smoking.
  Other Names: CBT
Drug: Bupropion — All medically eligible participants will be prescribed bupropion to begin 7 days before the quit date and continued through 12 weeks post-quit. Participants will be scheduled to begin at 150mg/day of bupropion for at least 3 days before titrating up to 300mg/day dose of bupropion.
  Other Names: Zyban
Behavioral: Cognitive Processing Therapy — 12 sessions of CPT, which is a well-established trauma-focused psychotherapy for PTSD that has demonstrated efficacy and effectiveness in Veterans.
  Other Names: CPT
Behavioral: Smoking Abstinence Reinforcement Therapy — Monetary reinforcement for smoking abstinence that is bioverified by breath carbon monoxide and saliva samples.
  Other Names: SMART
  Arms: CPT-SMART
Behavioral: Yoked Contingency Management — Participants in the yoked control will receive the monetary reinforcement of their yoked participant regardless of smoking abstinence or session attendance.
  Other Names: Control CM
  Arms: Combined Contact Yoked Control

SUMMARY:
Smoking is the leading cause of preventable illness, disability, and death in the United States. The rate of smoking is disproportionately higher among Veterans with posttraumatic stress disorder (PTSD). Unfortunately, smoking cessation efforts that are effective in the general population have shown limited effectiveness in smokers with PTSD. The high smoking rate and difficulty with achieving abstinence indicate a critical need to develop effective interventions for Veterans who smoke and have PTSD. The investigators' data indicate that negative emotions and trauma reminders are associated with relapse for smokers with PTSD. In this context, an ideal strategy may be to combine evidence-based PTSD treatment with intensive smoking cessation treatment to maximize quit rates.

Cognitive processing therapy (CPT) is a well-established evidence-based treatment for PTSD. The investigators have successfully developed a treatment manual that combines CPT with cognitive-behavioral counseling for smoking cessation. Contingency management (CM) is another intensive behavioral treatment that has been shown to help with reducing smoking. CM provides positive reinforcers such as money to individuals misusing substances contingent upon abstinence from use. The primary goal of this study is to evaluate the efficacy of a treatment that combines CM with cognitive-behavioral smoking cessation counseling, smoking cessation medication, and CPT. Proposed is a randomized, two-arm clinical trial in which 120 Veteran smokers with PTSD will be randomized to either: 1) COGNITIVE PROCESSING THERAPY with SMOKING ABSTINENCE REINFORCEMENT THERAPY (CPT-SMART) or 2) COMBINED CONTACT CONTROL, an intervention identical to CPT-SMART in PTSD and smoking treatment, except for using payment that is not contingent on abstinence.

Specific aims include: AIM 1) To evaluate the efficacy of CPT-SMART on rates of short- and long-term abstinence from cigarettes; AIM 2) To evaluate the impact of CPT-SMART on treatment engagement and utilization; and an EXPLORATORY AIM) To explore mechanisms of CPT-SMART on long-term smoking abstinence. The positive public health impact of reducing smoking among Veterans with PTSD could be enormous as it would prevent significant smoking-related morbidity and mortality.

DETAILED DESCRIPTION:
Smoking is the leading cause of preventable illness, disability, and death in the United States. The rate of smoking is disproportionately higher among Veterans with posttraumatic stress disorder (PTSD). Unfortunately, smoking cessation efforts that are effective in the general population have shown limited effectiveness in smokers with PTSD. The high smoking rate and difficulty with achieving abstinence indicate a critical need to develop effective interventions for PTSD smokers. The investigators' data indicate that negative affect and trauma reminders are a significant antecedent of relapse for PTSD smokers. Further, despite evidence that nicotine may exacerbate PTSD symptoms, many smokers with PTSD expect that smoking helps manage their symptoms. In this context, an ideal strategy may be to combine evidence-based PTSD treatment with intensive smoking cessation treatment to maximize quit rates in this at-risk population.

Cognitive processing therapy (CPT) is a well-established evidence-based treatment for PTSD. The investigators have successfully developed a treatment manual that integrates CPT with guideline-concordant cognitive-behavioral counseling for smoking cessation. Contingency management (CM) is an intensive behavioral treatment that has demonstrated efficacy for reducing smoking in a range of difficult-to-treat populations, including individuals with psychiatric disorders. CM provides positive reinforcers (e.g., vouchers, money) to individuals misusing substances contingent upon bioverified abstinence from drug use. The primary goal of the current study is to evaluate the efficacy of an intervention that combines clinic-based CM using twice weekly monitoring with salivary cotinine test strips, cognitive-behavioral smoking cessation counseling, smoking cessation medication, and evidence-based PTSD treatment. Proposed is a randomized, two-arm clinical trial in which 120 Veteran smokers with PTSD will be randomized to either: 1) COGNITIVE PROCESSING THERAPY with SMOKING ABSTINENCE REINFORCEMENT THERAPY (CPT-SMART) - an intervention that combines evidenced-based PTSD treatment with guideline-concordant cognitive-behavioral smoking cessation counseling, bupropion, and intensive behavioral therapy through CM; or 2) COMBINED CONTACT CONTROL: an intervention identical to CPT-SMART in PTSD and smoking treatment, except for using non-contingent payment (i.e., yoked CM) to control for compensation and monitoring.

Specific aims include: AIM 1) To evaluate the efficacy of CPT-SMART on rates of short- and long-term abstinence from cigarettes (assessed with multiple measures including bioverified abstinence) measured at 1-week post-treatment, 4-months, and 6 months; AIM 2) To evaluate the impact of CPT-SMART on treatment engagement and utilization; and an EXPLORATORY AIM) To explore mechanisms of CPT-SMART on long-term smoking abstinence, including self-efficacy, salience of smoking, and psychiatric symptom reduction. The VA has already implemented CM for treatment of substance abuse. If shown efficacious, a combined PTSD treatment plus incentive-based approaches for smoking could be implemented into specialty PTSD programs. The positive public health impact of reducing smoking among Veterans with PTSD could be enormous as it would prevent significant smoking-related morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Is Veteran
* Is between the ages of 18 and 80
* Smokes ten or more cigarettes per day for the past year
* Has been smoking for at least the past year
* Meets criteria for current PTSD
* Speaks and writes English
* Is willing to attempt smoking cessation and trauma-focused psychotherapy

Exclusion Criteria:

* Has had myocardial infarction in the past 6 months
* Uses other forms of nicotine that he/she is unwilling to stop
* Is pregnant
* Has a primary psychotic disorder
* Has a current substance use disorder other than tobacco use disorder
* Has a contraindication to bupropion use with no medical clearance to use it
* Is unwilling to use bupropion
* Is receiving other behavioral smoking counseling or trauma-focused therapy or plans to do so during the study period
* Is currently imprisoned or in psychiatric hospitalization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Number of participants whose self-report of 7 day point prevalence abstinence from smoking is bioverified | 6 month follow-up
  7-day point prevalence abstinence is defined as no smoking in the prior 7 days.

SECONDARY OUTCOMES:
Number of participants whose self-report of 30 day point prevalence abstinence from smoking is bioverified | 6 month follow-up
  30-day point prevalence abstinence is defined as no smoking in the prior 30 days.
Number of participants whose self-report of 7 day point prevalence abstinence from smoking is bioverified | 4 month follow-up
  7-day point prevalence abstinence is defined as no smoking in the prior 7 days.
Number of participants whose self-report of 30 day point prevalence abstinence from smoking is bioverified | 4 month follow-up
  30-day point prevalence abstinence is defined as no smoking in the prior 30 days.
Number of participants who self-report prolonged abstinence | 4 month follow-up
  Prolonged abstinence is defined as 30 days abstinent.
Number of participants who self-report prolonged abstinence | 6 month follow-up
  Prolonged abstinence is defined as 30 days abstinent.
Number of participants who self-report early abstinence | Measured at the post-treatment visit (2 weeks after treatment completed)
  Early abstinence is defined as 2 consecutive sessions abstinent in first month of quit attempt.
Number of participants who attended eight or more sessions of combined CPT and CBT for smoking | Measured at the post-treatment visit (2 weeks after treatment completed)
  Those who complete eight or more treatment sessions will be considered to have had an adequate treatment dose.
Number of sessions attended by participants | Measured at the post-treatment visit (2 weeks after treatment completed)
  The average number of treatment sessions attended by participants in each group will be considered a measure of treatment engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Dedert, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to attend individual participant data.

DOCUMENTS (1):
  • Informed Consent Form (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT03978442/ICF_000.pdf